CLINICAL TRIAL: NCT06124469
Title: Validation of The Ultrasound Neck Node Reporting and Data System (UNN-RADS) Scale for Diagnosing Lymph Node Metastasis in Patients With History of Thyroid Cancer
Brief Title: UNN-RADS Scale for Diagnosing Lymph Node Metastasis in Patients With History of Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Hilda Elizabeth Macías Cervantes, PhD, Instituto Mexicano del Seguro Social
Other Study IDs: 3
Record Dates: First submitted 2023-11-06; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Thyroid Cancer; Lymph Node
Keywords: Lymph node; Thyroid cancer; Ultrasonography; Metastasis
MeSH Terms: conditions — Thyroid Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 21 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Benign lymph nodes: Categories UNN-RADS 1 and 2 (test negative)
  Interventions: Diagnostic Test: US-guided fine needle aspiration (FNA)
- Metastatic lymph nodes: Categories UNN-RADS 3, 4, and 5 (test positive).
  Interventions: Diagnostic Test: US-guided fine needle aspiration (FNA)

INTERVENTIONS:
Diagnostic Test: US-guided fine needle aspiration (FNA) — This study enrolled consecutive patients in follow-up for DTC history who underwent US-guided fine needle aspiration (FNA) of the LNs for suspicious metastatic cervical

SUMMARY:
In 2020, Sarda-Inman et al., developed the Ultrasound Neck Node Reporting and Data System (UNN-RADS) scale that allows decision-making about when it is appropriate to perform FNA of a cervical lymph node, evaluating seven ultrasonographic descriptors (shape, margins, echogenicity, echogenicity of the hilum, vascularity and the presence/absence of calcifications, and cystic degeneration), features that have been associated with metastatic lymph nodes, with scores ranging from 0 to 3 points, which allows categorize into 5 different risk groups. Thus, the objective of this study is to evaluate the ultrasound characteristics of metastatic LN in patients undergoing TC follow-up and to validate the UNN-RADS scale for the diagnosis of LN Metastasis in Patients with a history of TC.

DETAILED DESCRIPTION:
This study enrolled consecutive patients in follow-up for differentiated thyroid cancer (DTC) history who underwent US-guided fine needle aspiration (FNA) of the LNs for suspicious metastatic cervical lymph nodes. Patients were included if they 1) had previous history of DTC, 2) both sexes with age over 18 years old, and 3) underwent FNA of the LNs for any suspected features corresponding with at least UNN-RADS 1. Patients were excluded if they underwent FNA of the LNs for persistent or recurrent disease after surgery for thyroid cancer, had previous bilateral cervical lymph node dissection as initial treatment, or the FNA results were not concluded.

UNN-RADS 1 y 2 and UNN-RADS 3, 4 and 5 were grouped for analysis purpose. Diagnostic performance of UNN-RADS scale were assessed in terms of sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV), positive likelihood ratios (+LR), negative likelihood ratios (-LR) and accuracy, as well as with a receiver operating characteristic (ROC) curve.

ELIGIBILITY:
Inclusion Criteria:

* 1) had previous history of DTC 2) both sexes with age over 18 years old 3) underwent FNA of the LNs for any suspected features corresponding with at least UNN-RADS 1

Exclusion Criteria:

* 1) underwent FNA of the LNs for persistent or recurrent disease after surgery for thyroid cancer 2) had previous bilateral cervical lymph node dissection as initial treatment 3) FNA results were not concluded

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients in follow-up for DTC history who underwent US-guided fine needle aspiration (FNA) of the LNs for suspicious metastatic cervical lymph nodes at Unidad Médica de Alta Especialidad HE 1 CMN Bajío
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
metastatic lymph node | All biopsy samples were sent to the pathology department of the unit, where final results were obtained in approximately 2-3 weeks.
  Fine needle aspiration biopsy (FNA) results were the gold standard (metastatic or benign).

CONTACTS AND LOCATIONS:
Overall Officials: Hilda Maciaqs, PhD, Study Chair — Instituto Mexicano del Seguro Social
Locations (1):
- Unidad Medica de Alta Especialidad No. 1, Bajío, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated or analyzed during the study are available from the principal investigator on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 month

REFERENCES:
- [Result] Ryu KH, Lee KH, Ryu J, Baek HJ, Kim SJ, Jung HK, Kim SM. Cervical Lymph Node Imaging Reporting and Data System for Ultrasound of Cervical Lymphadenopathy: A Pilot Study. AJR Am J Roentgenol. 2016 Jun;206(6):1286-91. doi: 10.2214/AJR.15.15381. Epub 2016 Apr 12. PMID 27070179
- [Result] Ahuja AT, Ying M. Sonographic evaluation of cervical lymph nodes. AJR Am J Roentgenol. 2005 May;184(5):1691-9. doi: 10.2214/ajr.184.5.01841691. PMID 15855141
- [Result] Prativadi R, Dahiya N, Kamaya A, Bhatt S. Chapter 5 Ultrasound Characteristics of Benign vs Malignant Cervical Lymph Nodes. Semin Ultrasound CT MR. 2017 Oct;38(5):506-515. doi: 10.1053/j.sult.2017.05.005. Epub 2017 May 20. PMID 29031367
- [Result] Ni X, Xu S, Zhan W, Zhou W. Ultrasonographic features of cervical lymph node metastases from medullary thyroid cancer: a retrospective study. BMC Med Imaging. 2022 Aug 29;22(1):151. doi: 10.1186/s12880-022-00882-7. PMID 36038830
- [Result] Meyer JE, Steffen A, Bienemann M, Hedderich J, Schulz U, Laudien M, Quetz J, Wollenberg B. Evaluation and development of a predictive model for ultrasound-guided investigation of neck metastases. Eur Arch Otorhinolaryngol. 2012 Jan;269(1):315-20. doi: 10.1007/s00405-011-1611-1. Epub 2011 May 6. PMID 21547389
- [Result] Sarda Inman ED, Valdez Rojas AM. Ultrasound Neck Node Reporting and Data System (UNN-RADS) for lymphadenopathy: A structured report. J Mex Fed Radiol Imaging 2022;3:151-163.